CLINICAL TRIAL: NCT05047796
Title: Effects of Osteopathic Visceral Manipulation on the Autonomic Nervous System, Balance and Gastrointestinal Disturbances in Individuals With Parkinson's Disease: a Randomized Clinical Trial
Brief Title: Effects of Osteopathic Visceral Manipulation on the Autonomic Nervous System, Balance and Gastrointestinal Disturbances in Individuals With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Docusse de Osteopatia e Terapia Manual (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18945219.4.0000.5402
Record Dates: First submitted 2021-09-03; First posted 2021-09-17 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Each participant will be randomly assigned to the intervention group or placebo group by an independent study evaluator. Data will be secretly allocated through sealed, opaque envelopes. After the randomization process, the participant will be evaluated by a researcher who will not have knowledge about the distribution of the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Protocol (Experimental): Visceral osteopathic techniques
  Interventions: Other: Intervention Protocol
- Sham Protocol (Sham Comparator): Simulated visceral osteopathic techniques
  Interventions: Other: Sham Protocol

INTERVENTIONS:
Other: Intervention Protocol — The intervention protocol will consist of visceral osteopathic techniques and will be performed by a professional who has 17 years of clinical experience in the field of Osteopathy.
  Arms: Intervention Protocol
Other: Sham Protocol — The sham protocol will be performed by a professional who has 17 years of clinical experience in the field of Osteopathy. The sham protocol will consist of simulation of therapy, where the therapist will place his hands in the same regions of the intervention protocol, without therapeutic intent
  Arms: Sham Protocol

SUMMARY:
Introduction: Parkinson's disease (PD) is responsible for several changes in the body, such as balance, gastrointestinal and autonomic disorders and are associated with impairments in the clinical prognosis of these individuals. In this sense, therapies capable of minimizing this impact are extremely important. Osteopathy has become an alternative treatment for individuals with neurological disorders and has been shown to be effective in treating various conditions, including PD. Objective: a) to evaluate the acute effect of visceral manipulation directed to the intestines and visceral plexuses in the autonomic nervous system of PD patients; b) identify the effect of this approach, after four visits, on balance, plantar pressure, gastrointestinal disorders and autonomic nervous system in this population. Materials and Methods: For this randomized clinical trial, 28 adults diagnosed with PD will be recruited. Subjects will be randomized to protocols in two groups: intervention protocol and placebo protocol, where both will consist of 4 visits twice a week. The intervention protocol will consist of osteopathic manipulative techniques and the sham protocol will consist of simulation of therapy, where the therapist will place his hands in the same regions of the intervention protocol, with superficial contact and without therapeutic intention in each region. The outcome measures of the study will consist of Berg balance assessment and plantar pressure, Rome survey on gastrointestinal disorders, and assessment of autonomic modulation by means of heart rate variability analysis. Volunteers and evaluators will be blind to the protocol and not informed of their order. Only the person responsible for the intervention will not be blind to the protocol. Data will be analyzed according to normality (Shapiro-Wilk test), and comparisons of outcomes between the moments (pre and post) will be performed using the T-student test for paired data or Wilcoxon, as normal and for comparisons between protocols. placebo and intervention, Student's T-test for unpaired data or Mann-Whitney test according to normality will be applied. The adopted statistical significance will be fixed at 5%.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's;
* Not having cardiorespiratory diseases;
* Not being a smoker;
* Do not use alcoholic beverages;
* No cognitive deficit;
* No osteoarticular deformities, plantar ulcers, total or partial amputation of the feet;
* They do not need auxiliary devices for walking

Exclusion Criteria:

* Data from individuals with a series of heart rate intervals with less than 95% of sinus beats will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Change in heart rate variability | T0= before the protocol (15 minutes); T1= until 48 hours after the end protocol (15 minutes)
  For the analysis, frequency domain indices (LF, HF, LF/HF), time domain (SDNN, RMSSD) and geometric indices will be used

SECONDARY OUTCOMES:
Change in balance | T0= before the protocol; T1= until 48 hours after the end protocol
  For balance analysis we will use the Berg balance scale, validated for the Brazilian population. The overall score is 56 points. A score from 0 to 20 represents impairment of balance, 21 to 40 is acceptable balance, and 41-56 is good balance.
Change in plantar pressure | T0= before the protocol; T1= until 48 hours after the end protocol
  The static plantar pressure profile will be obtained through pressure sensors present in the platform

CONTACTS AND LOCATIONS:
Locations (1):
- Anne Kastelianne, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared for any researcher that requests the data by electronic address
Supporting Information: Study Protocol, SAP
Time Frame: After one year of publication
Access Criteria: To receive the data, the researcher must have sent a request to nupi@idot.com.br